CLINICAL TRIAL: NCT00243932
Title: Clinical Trial of High Dose CoQ10 in ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAA1536; R01NS048125 (NIH)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Results first posted 2011-03-17 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Amyotrophic Lateral Sclerosis; Lou Gehrig's Disease
Keywords: amyotrophic lateral sclerosis; ALS; Lou Gehrig's disease; CoQ10; coenzyme Q10; antioxidants; free radicals; mitochondrial dysfunction
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Mitochondrial Diseases | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2,700 mg CoQ10 (Experimental)
  Interventions: Drug: coenzyme Q10
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 1,800 mg CoQ10 (Experimental)
  Interventions: Drug: coenzyme Q10

INTERVENTIONS:
Drug: coenzyme Q10 — antioxidant and mitochondrial cofactor, given in capsules three times daily
  Other Names: Coenzyme Q 10; CoQ10
  Arms: 1,800 mg CoQ10; 2,700 mg CoQ10
Drug: Placebo — Placebo capsules, indistinguishable from CoQ10 capsules, given three times daily
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the efficacy and preferred dose of CoQ10 in individuals with ALS for a possible future phase III study.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive and devastating neurodegenerative disorder. Available treatment for ALS remains scarce. Oxidative stress and mitochondrial dysfunction have been implicated in the pathophysiology of ALS. Oxidative stress refers to the effects of cell-damaging reactive oxygen species, also known as free radicals. Oxidative stress is thought to contribute to nerve cell loss in ALS. Mitochondria are organelles within each cell that are sometimes called "powerhouses of the cell" because cellular energy metabolism is located within the mitochondria.

Coenzyme Q10 (CoQ10), a mitochondrial cofactor known for its antioxidant properties, has prolonged survival in the mouse model of ALS and has slowed functional decline in another neurodegenerative disorder, Parkinson's disease. The goals of this double-blind, placebo-controlled, two-dose comparison phase II study are to obtain preliminary efficacy data and to select the preferred dose for a larger phase III study.

Participants were randomly assigned to CoQ10 (at two different dose levels) or placebo in the first stage, then the 2,700 mg dose was selected in the second stage. Duration of the trial was 9 months with a total of 7 visits.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of definite, probable, or laboratory-supported probable ALS
* Negative pregnancy test for women of childbearing age and adequate birth control measures
* Subjects must be able and willing to give informed consent and must be capable of complying with the trial procedures
* Forced Vital Capacity (FVC) >/= 60% of predicted
* Age 21 to 85 years, inclusive
* Disease duration of less than 5 years
* Subjects may take riluzole (without change in dose for more than 30 days before enrollment)
* Patients who have taken CoQ10 in the past will be eligible if they stop at least 30 days before enrollment
* Patients who have taken vitamin E in the past will be eligible if they stop at least 14 days before enrollment

Exclusion Criteria:

* Dependency on mechanical ventilation (non-invasive ventilation > 23 hours)
* Severe and unstable concomitant medical or psychiatric illness
* Insufficiently controlled diabetes mellitus
* Concomitant warfarin therapy
* Women who are breast feeding or have a high likelihood of pregnancy
* Significant hepatic dysfunction
* Forced Vital Capacity (FVC) less than 60%
* Exposure to CoQ10 within 30 days of enrollment
* Exposure to other experimental medications within 30 days of enrollment
* Exposure to vitamin E within 14 days of enrollment
* Sensitivity to color additive FD&C Yellow No. 5
* Sensitivity to aspirin

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2005-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petra Kaufmann, MD, Principal Investigator — Assistant Professor, Division of Neuromuscular Disease, Columbia University Medical Center (Clinical Principal Investigator); J. L. P. Thompson, Ph.D., Principal Investigator — Director, Statistical Analysis Center, Department of Biostatistics, Mailman School of Public Health (Statistical Principal Investigator); Hiroshi Mitsumoto, Principal Investigator — Wesley J. Howe Professor of Neurology at the New York Presbyterian Hospital/Columbia University Medical Center
Locations (19):
- United States (19):
  - University of Arkansas for Medical Sciences, Department of Neurology, Little Rock, Arkansas
  - California Pacific Medical Center, San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - University of Colorado Health Sciences, Dept of Neurology, Denver, Colorado
  - Yale University School of Medicine, Department of Neurology, New Haven, Connecticut
  - Northwestern University, Department of Neurology,, Chicago, Illinois
  - University of Chicago, Department of Neurology, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Dept of Neurology, College of Medicine, Lexington, Kentucky
  - Brigham and Women's Hospital , Department of Neurology, Boston, Massachusetts
  - Baystate Medical Center, Division of Critical Care Research, Springfield, Massachusetts
  - Minneapolis Medical Research Foundation, ,, Minneapolis, Minnesota
  - Washington University in St. Louis School of Medicine, Department of Neurology, St Louis, Missouri
  - Columbia Presbyterian Medical Center, The Neurological Institute, New York, New York
  - State University of New York Upstate Medical, Neurology Department, Syracuse, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Drexel University, Dept of Neurology, Philadelphia, Pennsylvania
  - University of Texas, Health Science Center at San Antonio, Division of Neurology, San Antonio, Texas
  - University of Vermont, Neurology Department, Burlington, Vermont

REFERENCES:
- [Result] Kaufmann P, Thompson JL, Levy G, Buchsbaum R, Shefner J, Krivickas LS, Katz J, Rollins Y, Barohn RJ, Jackson CE, Tiryaki E, Lomen-Hoerth C, Armon C, Tandan R, Rudnicki SA, Rezania K, Sufit R, Pestronk A, Novella SP, Heiman-Patterson T, Kasarskis EJ, Pioro EP, Montes J, Arbing R, Vecchio D, Barsdorf A, Mitsumoto H, Levin B; QALS Study Group. Phase II trial of CoQ10 for ALS finds insufficient evidence to justify phase III. Ann Neurol. 2009 Aug;66(2):235-44. doi: 10.1002/ana.21743. PMID 19743457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized between April, 2005 and May, 2007. The last participant completed the trial March 2008.
Pre-assignment Details: Exclusion criteria were forced vital capacity (FVC) of less than 60%, severe medical illness, or disease onset more than 5 years before study entry.
Groups:
- 2700mg CoQ10: 35 subjects from stage 1 + 40 new subjects; all taking 2,700mg CoQ10 - total 75.
- Placebo: 35 subjects from stage 1 + 40 new subjects; all receiving placebo - total 75.
- 1,800 mg CoQ10: 35 patients. This dose group was discontinued after stage 1; only the 2,700 mg group was compared with placebo in the efficacy analysis.
Period: Stage 1: Dose Selection
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10
Started | 35 | 35 | 35
Completed | 33 | 35 | 35
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: Stage 2: Efficacy
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10
Started | 40 (40 newly randomized pts. Efficacy analysis included Stage 1 + Stage 2 patients) | 40 (40 newly randomized pts. Efficacy analysis included Stage 1 + Stage 2 patients) | 0 (No new pts. randomized because selection procedure in Stage 1 selected the 2,700 mg dose.)
Completed | 40 | 40 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10 | Total
Number analyzed (Participants) | 75 | 75 | 35 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 62 | 62 | 23 | 147
  >=65 years | 13 | 13 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10.8) | 56.9 (11) | 58.9 (12.5) | 56.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 10 | 74
  Male | 40 | 46 | 25 | 111
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 35 | 185

OUTCOME MEASURES:

1. Primary Outcome: Change in the ALS Functional Rating Scale-revised (ALSFRSr) Score.
Description: The ALSFRSr, a questionnaire-based scale assessing daily living function ranging from 48 (best score) to 0 (worst), was administered to the patient, or to a proxy if the patient could not communicate effectively. Decline was defined as ALSFRSr at baseline minus ALSFRSr at month 9. Thus a positive value indicates worsening.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 2700mg CoQ10: 40 new subjects and 35 subjects from stage 1 all taking 2,700mg CoQ10 - total 75.
  Stage 1 - 35 participants per group compared CoQ10 doses of 1,800mg and 2,700 mg/day and placebo.
- Placebo: 40 new subjects plus 35 subjects from stage 1 receiving placebo - total 75.
- 1,800 mg CoQ10: 35 patients. Mean and SD are presented but this group was not included in the efficacy analysis because the 1,800 mg dose was discontinued after stage 1.
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10
Number analyzed (Participants) | 73 | 75 | 35
units on a scale | 8.80 (7.34) | 9.44 (8.82) | 10.9 (9.3)
Statistical Analysis 1: Comparison: 2700mg CoQ10 vs Placebo; Null hypothesis: 2,700mg CoQ10 is at least 20% superior to placebo; Test type: Superiority or Other; p = 0.14, futility (non-superiority)

2. Secondary Outcome: Change in Fatigue Severity Scale
Description: The change over 9 months in fatigue severity scale. A 9-item scale measuring the impact of fatigue. Scores range from 7 (strongly disagree)-63 (strongly agree) with higher scores indicating a worse outcome.
Time Frame: 9 months
Population: 1,800 mg CoQ10 group was not included in the efficacy analysis because the 1,800 mg dose was discontinued after stage 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 1,800 mg CoQ10: 1,800 mg CoQ10 (35 patients). This group was not included in the efficacy analysis because the 1,800 mg dose was discontinued after stage 1.
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10
Number analyzed (Participants) | 75 | 75 | 0
score on a scale | 0.71 (1.21) | 0.88 (1.51) |

3. Secondary Outcome: Change in Forced Vital Capacity
Description: The change over 9 months in forced vital capacity is the volume (liters) of gas that can be exhaled by maximum voluntary effort following deep inspiration. The best of three trials will be recorded. The result is recorded as percentage of predicted for age, height and weight.
Time Frame: 9 months
Population: 1,800 mg CoQ10 group was not included in the efficacy analysis because the 1,800 mg dose was discontinued after stage 1.
Measure: Mean (Standard Deviation); unit: Percent of Predicted
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10
Number analyzed (Participants) | 75 | 75 | 0
Percent of Predicted | 0.20 (0.15) | 0.17 (0.18) |

4. Secondary Outcome: Change in Short Form (SF)-36 Score (Physical)
Description: The change over 9 months in SF-36 score, which is a quality of life measure. Scores range from 0-100 with a higher score indicating a better outcome.
Time Frame: 9 months
Population: 1,800 mg CoQ10 group was not included in the efficacy analysis because the 1,800 mg dose was discontinued after stage 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10
Number analyzed (Participants) | 75 | 75 | 0
score on a scale | 4.22 (8.02) | 6.04 (6.85) |

5. Secondary Outcome: Change in Short Form (SF)-36 Score (Mental)
Description: as for outcome 4
Time Frame: 9 months
Population: 1,800 mg CoQ10 group was not included in the efficacy analysis because the 1,800 mg dose was discontinued after stage 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10
Number analyzed (Participants) | 75 | 75 | 0
score on a scale | 2.87 (11.78) | 5.01 (11.69) |

ADVERSE EVENTS:
Arm/Group | 2700mg CoQ10 | Placebo | 1,800 mg CoQ10
Serious Adverse Events (participants affected / at risk) | 18/75 | 19/75 | 10/35
Other Adverse Events (participants affected / at risk) | 63/75 | 64/75 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2700mg CoQ10 (N=75) | Placebo (N=75) | 1,800 mg CoQ10 (N=35)
Peg placement (Surgical and medical procedures) | 5 (5) | 4 (4) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3) | 1 (1)
Pain (General disorders) | 3 (4) | 0 (0) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Other (General disorders) | 14 (16) | 9 (9) | 1 (2)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GI (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2700mg CoQ10 (N=75) | Placebo (N=75) | 1,800 mg CoQ10 (N=35)
Neurology - Other (Nervous system disorders) | 29 (68) | 18 (40) | 8 (16)
Pain (General disorders) | 21 (42) | 20 (21) | 10 (14)
Nausea (Gastrointestinal disorders) | 13 (18) | 16 (19) | 4 (4)
Constipation (Gastrointestinal disorders) | 17 (19) | 10 (10) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 18 (22) | 6 (8)
Mood alteration (Psychiatric disorders) | 15 (20) | 7 (8) | 7 (7)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 11 (15) | 6 (6)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 10 (13) | 6 (6) | 5 (5)
BIPAP/NIPPV (Surgical and medical procedures) | 8 (8) | 6 (6) | 3 (3)
Gastrointestinal - Other (Gastrointestinal disorders) | 8 (11) | 6 (6) | 5 (5)
Edema: limb (Cardiac disorders) | 8 (12) | 5 (5) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 6 (8) | 6 (8) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 6 (7) | 5 (5) | 2 (2)
Infection with unknown ANC (Infections and infestations) | 5 (6) | 6 (8) | 0 (0)
Other (General disorders) | 50 (244) | 51 (231) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No